CLINICAL TRIAL: NCT01738503
Title: Open-Label, Multicenter, Multiple Dose Study of Safety, Tolerability, Pharmacokinetics, Efficacy Markers, and Opioid Receptor Availability of Subcutaneous Injections of Depot Buprenorphine in Treatment Seeking Opioid-Dependent Subjects
Brief Title: Multiple Dose Pharmacokinetics Depot Buprenorphine in Opioid-Dependent Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RB-US-12-0005
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-01

CONDITIONS: Opioid Related Disorder
Keywords: Opioid Dependence, Buprenorphine, Depot, SUBUTEX, RBP-6000
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- (8 mg) RBP-6000: 50 mg (Experimental): Participants are stabilized by day -5 on Subutex 8 mg. During the study, four subcutaneous (SC) injections containing RBP-6000 50 mg are given at 28 day intervals.
  Interventions: Drug: RBP-6000; Drug: Subutex
- (12 mg) RBP-6000: 100 mg (Experimental): Participants are stabilized by day -5 on Subutex 12 mg. During the study, four subcutaneous (SC) injections containing RBP-6000 100 mg are given at 28 day intervals
  Interventions: Drug: RBP-6000; Drug: Subutex
- (24 mg) RBP-6000: 200 mg (Experimental): Participants are stabilized by day -5 on Subutex 24 mg. During the study, four subcutaneous (SC) injections containing RBP-6000 200 mg are given at 28 day intervals.
  Participants who receive RBP-6000 containing 200 mg buprenorphine and reach Day 112 (and have received all 4 planned SC injections) have the option to participate in the Positron Emission Tomography (PET) Pilot substudy. In the PET Pilot sub-study participants remain on 200 mg SC injections at 28 day intervals for an additional 6-9 intervals until they complete an magnetic resonance imaging (MRI) and a PET scan and pharmacokinetic samples at week 1 and week 4 post injection.
  Interventions: Drug: RBP-6000; Drug: Subutex
- (8 mg) RBP-6000: 100 mg (Experimental): Participants are stabilized by day -5 on Subutex 8 mg. During the study, four subcutaneous (SC) injections containing RBP-6000 100 mg are given at 28 day intervals.
  Interventions: Drug: RBP-6000; Drug: Subutex
- (14 mg) RBP-6000: 200 mg (Experimental): Participants are stabilized by day -5 on Subutex 14 mg. During the study, four subcutaneous (SC) injections containing RBP-6000 200 mg are given at 28 day intervals.
  Participants who receive RBP-6000 containing 200 mg buprenorphine and reach Day 112 (and have received all 4 planned SC injections) have the option to participate in the Positron Emission Tomography (PET) Pilot substudy. In the PET Pilot sub-study participants remain on 200 mg SC injections at 28 day intervals for an additional 6-9 intervals until they complete an magnetic resonance imaging (MRI) and a PET scan and pharmacokinetic samples at week 1 and week 4 post injection.
  Interventions: Drug: RBP-6000; Drug: Subutex
- (8-24 mg) RBP-6000: 300 mg (Experimental): Participants are stabilized by day -5 on a Subutex between 8-24 mg. During the study, four subcutaneous (SC) injections containing RBP-6000 300 mg are given at 28 day intervals.
  Interventions: Drug: RBP-6000; Drug: Subutex

INTERVENTIONS:
Drug: RBP-6000 — 18% Buprenorphine Sterile Solution for subcutaneous (SC) injection using the ATRIGEL® Delivery System. Each injection of RBP-6000 is separated by a minimum of 28 days and given on alternate sides of the participant's abdomen.
  Other Names: buprenorphine
Drug: Subutex — Participants were inducted and stabilized over a 14-day period (study days -14 to -1) on SUBUTEX sublingual tablets. Tablets are placed under the tongue until dissolved.
  Other Names: buprenorphine

SUMMARY:
This is an open-label study in treatment seeking opioid-dependent subjects for safety, tolerability, pharmacokinetics (PK), efficacy markers, and opioid receptor availability of subcutaneous injections of depot buprenorphine after induction and stabilization of treatment seeking subjects onto Subutex.

Subjects were planned to receive 4 subcutaneous (SC) injections of RBP-6000 separated by 28 days (Cohorts 1-5) or 6 SC injections of RBP-6000 separated by 28 days (Cohort 6) after a 13-day induction and dose stabilisation period on SUBUTEX Sublingual (SL) tablet at dose levels of 8-24 mg.

DETAILED DESCRIPTION:
* Open-label SUBUTEX Sublingual Tablet Induction and Stabilisation Period After completing the screening period, subjects entered an open-label SUBUTEX SL tablet induction and stabilisation period to achieve stable daily doses of 8 mg, 12 mg, 14 mg, 24 mg or 8 - 24 mg (variable) during a 13 day inpatient (Day -14 to Day -1) period.
* Open-label Treatment Phase On Day 1, eligible subjects discontinued use of SUBUTEX SL tablet and received a subcutaneous (SC) injection of RBP-6000. The dose of RBP-6000 received and the cohort to which a subject was assigned depended upon the SUBUTEX SL tablet dose on Day -1.

  * Injection 1 (Day 1): 3 days inpatient post-dose (Day 1 to Day 3) and outpatient visits (Day 4 to Day 28); serial pharmacokinetic (PK) samples
  * Injection 2 (Day 29): 60-hour inpatient pre-dose and post-dose (Day 28 to Day 31) and outpatient visits (Day 32 to Day 56); sparse PK samples
  * Injection 3 (Day 57): 60-hour inpatient pre-dose and post-dose (Day 56 to Day 59) and outpatient visits (Day 60 to Day 84); sparse PK samples
  * Injection 4 (Day 85): 60-hour inpatient pre-dose and post-dose (Day 84 to Day 87) and outpatient visits (Day 88 to Day 113 [or Day 112 for Cohort 6]); serial PK samples
  * Cohort 6 ONLY: Injection 5 (Day 113): 60-hour inpatient pre-dose and post-dose (Day 112 to Day 115) and outpatient visits (Day 116 to Day 140); serial PK samples
  * Cohort 6 ONLY: Injection 6 (Day 141): 60-hour inpatient pre- and post-dose (Day 140 to Day 143) and outpatient visits (Day 144 to Day 169); serial PK samples
  * Safety Follow-up: weekly visits up to 60 days post-Injection 4 (PK Day 114 to Day 141) for subjects in Cohorts 1-5 who did not take part in the positron emission tomography (PET) imaging sub-study and up to 60 days post-Injection 6 (PK Day 169 to Day 197) for subjects in Cohort 6

The objective of the PET imaging sub-study was to evaluate the relationship between buprenorphine plasma levels and the ability of the 200 mg and 300 mg doses of RBP-6000 to reduce mu-opioid receptor availability measured with [11C]carfentanil and positron emission tomography (PET) scans. This objective was exploratory in nature and results are not reported as part of these summary results.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects
* Agree not to take any buprenorphine products other than those administered for the current study throughout participation in the study
* Body mass index (BMI) of >18.0 to < 33.0 kg/m

Exclusion Criteria:

* Participants with a current diagnosis requiring chronic opioid treatment
* Participants with a history of risk factors of Torsades de Pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome) or an ECG demonstrating a Fridericia's corrected QT interval (QTcF) >450 msec in males and QTcF > 470 in females at screening
* Abuse of buprenorphine or use of buprenorphine within 14 days of informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley D Vince, DO, Principal Investigator — Vince and Associates Clinical Research
Locations (1):
- Vince and Associates Clinical Research, Overland Park, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 395 subjects provided informed consent to participate in the main study and underwent screening procedures. Of these 395 subjects, 124 received study treatment.
Groups:
- SUBUTEX: Participants who entered the Induction/Stabalization period, were treated with SUBUTEX SL. Those who did not complete this period, did not continue into the Treatment period.
- Group 1 (8 mg) RBP-6000: 50 mg: Participants are stabilized by day -5 on Subutex 8 mg. During the study, four subcutaneous (SC) injections containing RBP-6000 50 mg are given at 28 day intervals.
- Group 2 (12 mg) RBP-6000: 100 mg: Participants are stabilized by day -5 on Subutex 12 mg. During the study, four subcutaneous (SC) injections containing RBP-6000 100 mg are given at 28 day intervals.
- Group 3 (24 mg) RBP-6000: 200 mg: Participants are stabilized by day -5 on Subutex 24 mg. During the study, four subcutaneous (SC) injections containing RBP-6000 200 mg are given at 28 day intervals.
  Participants who reach Day 113 (and have received all 4 planned SC injections) have the option to participate in the Positron Emission Tomography (PET) Pilot substudy. In the PET Pilot sub-study participants remain on 200 mg SC injections at 28 day intervals for an additional 6-9 intervals until they complete an magnetic resonance imaging (MRI) and a PET scan and pharmacokinetic samples at week 1 and week 4 post injection.
- Group 4 (8 mg) RBP-6000: 100 mg: Participants are stabilized by day -5 on Subutex 8 mg. During the study, four subcutaneous (SC) injections containing RBP-6000 100 mg are given at 28 day intervals.
- Group 5 (14 mg) RBP-6000: 200 mg: Participants are stabilized by day -5 on Subutex 14 mg. During the study, four subcutaneous (SC) injections containing RBP-6000 200 mg are given at 28 day intervals.
  Participants who reach Day 113 (and have received all 4 planned SC injections) have the option to participate in the Positron Emission Tomography (PET) Pilot substudy. In the PET Pilot sub-study participants remain on 200 mg SC injections at 28 day intervals for an additional 6-9 intervals until they complete an magnetic resonance imaging (MRI) and a PET scan and pharmacokinetic samples at week 1 and week 4 post injection.
- Group 6 (8-24 mg) RBP-6000: 300 mg: Participants are stabilized by day -5 on a Subutex between 8-24 mg. During the study, up to six subcutaneous (SC) injections containing RBP-6000 300 mg are given at 28 day intervals.
  Participants who reach Day 168 (and have received all 6 planned SC injections) have the option to participate in the Positron Emission Tomography (PET) Pilot substudy. In the PET Pilot sub-study participants remain on 300 mg SC injections at 28 day intervals for an additional 6 intervals until they complete an magnetic resonance imaging (MRI) and a PET scan and pharmacokinetic samples at week 1 and week 4 post injection.
Period: Induction/Stabilization (Days -14 to -1)
Arm/Group | SUBUTEX | Group 1 (8 mg) RBP-6000: 50 mg | Group 2 (12 mg) RBP-6000: 100 mg | Group 3 (24 mg) RBP-6000: 200 mg | Group 4 (8 mg) RBP-6000: 100 mg | Group 5 (14 mg) RBP-6000: 200 mg | Group 6 (8-24 mg) RBP-6000: 300 mg
Started | 124 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 89 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 35 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 35 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period
Arm/Group | SUBUTEX | Group 1 (8 mg) RBP-6000: 50 mg | Group 2 (12 mg) RBP-6000: 100 mg | Group 3 (24 mg) RBP-6000: 200 mg | Group 4 (8 mg) RBP-6000: 100 mg | Group 5 (14 mg) RBP-6000: 200 mg | Group 6 (8-24 mg) RBP-6000: 300 mg
Started | 0 | 15 | 15 | 15 | 15 | 15 | 14
Completed | 0 | 10 (Completed to Day 113 (4 injections)) | 10 (Completed to Day 113 (4 injections)) | 9 (Completed to Day 113 (4 injections)) | 7 (Completed to Day 113 (4 injections)) | 9 (Completed to Day 113 (4 injections)) | 6 (Completed to Day 113 (4 injections))
Not Completed | 0 | 5 | 5 | 6 | 8 | 6 | 8
Not completed — Adverse Event | 0 | 1 | 0 | 1 | 2 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 3 | 4 | 1 | 1 | 5
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 1 | 1 | 1
Not completed — Protocol Violation | 0 | 3 | 1 | 0 | 4 | 2 | 0
Not completed — Other | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: PET Imaging Sub-study
Arm/Group | SUBUTEX | Group 1 (8 mg) RBP-6000: 50 mg | Group 2 (12 mg) RBP-6000: 100 mg | Group 3 (24 mg) RBP-6000: 200 mg | Group 4 (8 mg) RBP-6000: 100 mg | Group 5 (14 mg) RBP-6000: 200 mg | Group 6 (8-24 mg) RBP-6000: 300 mg
Started | 0 | 0 | 0 | 0 | 0 | 3 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 1 (Completion defined as a total of 12 injections plus all PET images) | 1 (Completion defined as a total of 6 injections plus all PET images)
Not Completed | 0 | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Scheduling issues with imaging facility | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (8 mg) RBP-6000: 50 mg | Group 2 (12 mg) RBP-6000: 100 mg | Group 3 (24 mg) RBP-6000: 200 mg | Group 4 (8 mg) RBP-6000: 100 mg | Group 5 (14 mg) RBP-6000: 200 mg | Group 6 (8-24 mg) RBP-6000: 300 mg | Total
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 14 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (11.36) | 31.1 (11.14) | 30.1 (11.21) | 36.1 (14.87) | 36.2 (12.85) | 32.9 (11.00) | 33.8 (12.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 5 | 6 | 6 | 4 | 29
  Male | 12 | 10 | 10 | 9 | 9 | 10 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 3 | 3 | 5 | 5 | 3 | 26
  White | 8 | 11 | 12 | 10 | 10 | 11 | 62
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1 | 1 | 1 | 4
  Not Hispanic or Latino | 15 | 14 | 15 | 14 | 14 | 13 | 85
Weight [Mean (Standard Deviation); unit: kg] | 71.12 (12.929) | 73.71 (10.411) | 68.08 (9.900) | 74.43 (15.995) | 73.16 (12.753) | 74.64 (16.825) | 72.50 (13.159)
Height [Mean (Standard Deviation); unit: cm] | 173.41 (8.514) | 172.87 (8.532) | 170.50 (11.738) | 171.17 (8.701) | 168.71 (10.963) | 170.64 (11.469) | 171.22 (9.906)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 23.55 (3.084) | 24.67 (3.239) | 23.39 (2.298) | 25.26 (4.295) | 25.67 (3.635) | 25.36 (3.355) | 24.64 (3.394)
Other Opioid Use [Mean (Standard Deviation); unit: years] — Population: Missing participants reported no use
  years
    number analyzed (Participants) | 12 | 11 | 12 | 11 | 11 | 10 | 67
    (all) | 6.75 (5.545) | 6.18 (4.191) | 4.17 (2.887) | 5.27 (3.927) | 8.36 (9.770) | 6.30 (8.693) | 6.15 (6.165)
Heroin Use [Mean (Standard Deviation); unit: years] — Population: Missing participants reported no use
  years
    number analyzed (Participants) | 12 | 9 | 11 | 14 | 10 | 9 | 65
    (all) | 11.25 (10.463) | 9.78 (11.454) | 5.00 (5.604) | 11.64 (12.549) | 10.70 (7.987) | 8.56 (12.471) | 9.62 (10.292)
Smoking History (Nicotine Use) [Mean (Standard Deviation); unit: years] — Population: Missing participants reported no use
  years
    number analyzed (Participants) | 14 | 14 | 14 | 12 | 14 | 13 | 81
    (all) | 15.14 (10.596) | 10.64 (5.387) | 9.57 (8.225) | 19.83 (14.282) | 20.07 (11.526) | 17.31 (13.054) | 15.30 (11.243)

OUTCOME MEASURES:

1. Primary Outcome: Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: TEAE=any untoward medical occurrence that develops or worsens in severity after dispensation of the study drug and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator on a scale of mild, moderate and severe, with severe= a marked limitation in activity. Relation of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent one of the outcomes listed in this definition. A serious AE (SAE) is defined as any AE occurring at any dose that results in any of the following outcomes: death; lifethreatening AE; hospitalization or prolongation of existing hospitalization; a persistent or significant disability/incapacit
Time Frame: Days -14 to -1 (Subutex treatment), Days 1-316 (RBP-6000 treatment)
Population: Safety analysis group
Measure: Count of Participants; unit: Participants
Groups:
- SUBUTEX Only: Participants who entered the Induction/Stabalization period, were treated with SUBUTEX SL and did not continue into the Treatment period.
Arm/Group | SUBUTEX Only | Group 1 (8 mg) RBP-6000: 50 mg | Group 2 (12 mg) RBP-6000: 100 mg | Group 3 (24 mg) RBP-6000: 200 mg | Group 4 (8 mg) RBP-6000: 100 mg | Group 5 (14 mg) RBP-6000: 200 mg | Group 6 (8-24 mg) RBP-6000: 300 mg
Number analyzed (Participants) | 35 | 15 | 15 | 15 | 15 | 15 | 14
Participants
  >=1 TEAE | 24 | 15 | 15 | 15 | 15 | 15 | 14
  >=1 TEAE related to study drug | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=1 Severe TEAE | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Deaths | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=1 SAE other than death | 0 | 0 | 2 | 1 | 1 | 2 | 0
  Withdrew from study due to a TEAE | 0 | 1 | 0 | 1 | 2 | 2 | 2

2. Primary Outcome: Buprenorphine PK: % Fluctuation
Description: % Fluctuation was defined as the degree of fluctuation of buprenorphine plasma concentrations calculated as (Cmax-Cmin)/Cavg*100, expressed as a percentage. Cmax=maximum plasma concentration Cmin=minimum plasma concentration Cavg = average plasma concentration
  Results are reported across three timeframes:
  * Sublingual Period (Day -1 dose of SUBUTEX): a steady-state reading.
  * Plateau Parameters (Days 3-29 relative to RBP-6000 injections 1, 4 and 6)
  * Overall Parameters (Days 1-29 relative to RBP-6000 injections 1, 4 and 6)
  The PK sampling schedule was
  * hour 0 (predose) on days -7 to -1,
  * hours 0.5, 1,2,4,6, 8,12, 24 post-dose on Day -1
  * hours 0 (pre-dose) 1, 2, 4, 6, 8, 12, 20, 24, 25, 26, 28, 30, 32, 36, 44, 48, 144, 192, 240, 312, 384, 456, 528, 600, 672 post injections 1 and 4
  * hours 0 (pre-dose) 1, 2, 4, 6, 8, 12, 20, 24, 25, 26, 28, 30, 32, 36, 44, 48, 144, 192, 240, 312, 384, 456, 528, 600, 672, 846, 1008, 1200, 1344 post injection 6
Time Frame: Day -1, Days 1-29, 85-113, 141-197
Population: The PK analysis population was defined as any subject in Groups 1 - 6 who received a dose of RBP-6000 or at least 1 dose of SUBUTEX SL tablet and had an adequate number of PK samples collected to derive PK parameters.
Measure: Mean (Standard Deviation); unit: % of average concentration
Arm/Group | Group 1 (8 mg) RBP-6000: 50 mg | Group 2 (12 mg) RBP-6000: 100 mg | Group 3 (24 mg) RBP-6000: 200 mg | Group 4 (8 mg) RBP-6000: 100 mg | Group 5 (14 mg) RBP-6000: 200 mg | Group 6 (8-24 mg) RBP-6000: 300 mg
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 14
% of average concentration
  Sublingual Period | 256.993 (68.4944) | 272.702 (62.1424) | 233.978 (84.1776) | 268.690 (54.5116) | 227.874 (69.1437) | 245.513 (61.2524)
  Plateau: Injection 1: number analyzed (Participants) | 11 | 14 | 14 | 9 | 13 | 10
  Plateau: Injection 1 | 213.664 (50.7221) | 175.068 (69.0037) | 168.963 (31.8302) | 140.924 (39.3779) | 135.433 (31.4609) | 107.909 (33.9246)
  Plateau: Injection 4: number analyzed (Participants) | 10 | 12 | 10 | 9 | 10 | 5
  Plateau: Injection 4 | 68.333 (16.8729) | 63.611 (27.6839) | 42.699 (5.6645) | 41.275 (14.1786) | 47.282 (21.0395) | 53.383 (20.9467)
  Plateau: Injection 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1
  Plateau: Injection 6 |  |  |  |  | 22.597 | 31.376
  Overall: Injection 1: number analyzed (Participants) | 15 | 14 | 13 | 14 | 14 | 11
  Overall: Injection 1 | 315.777 (106.6237) | 234.098 (60.7481) | 234.598 (66.4979) | 213.254 (68.1754) | 206.691 (79.9858) | 220.854 (70.3346)
  Overall: Injection 4: number analyzed (Participants) | 10 | 11 | 9 | 8 | 7 | 2
  Overall: Injection 4 | 152.755 (75.3194) | 95.140 (20.9504) | 75.633 (17.3765) | 77.067 (21.4559) | 75.202 (28.4598) | 83.695 (12.8165)
  Overall: Injection 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0
  Overall: Injection 6 |  |  |  |  | 54.789 (1.6355) |

3. Primary Outcome: Buprenorphine PK: Area Under Plasma Concentration Time Curves (AUC)
Description: AUC calculated using the linear trapezoidal rule and requiring a minimum of 5 data points for each time range.
  Results are reported across four timeframes:
  * Sublingual Period (Day -1 dose of SUBUTEX): a steady-state reading at hours 0-24.
  * Initial Burst Parameters (Days 1-2 relative to RBP-6000 injections 1, 4 and 6) at hours 0-48
  * Plateau Parameters (Days 3-29 relative to RBP-6000 injections 1, 4 and 6) at hours 48-672
  * Overall Parameters (Days 1-29 relative to RBP-6000 injections 1, 4 and 6) at hours 0-24, hours 0-672
  The PK sampling schedule was
  * hour 0 (predose) on days -7 to -1,
  * hours 0.5, 1,2,4,6, 8,12, 24 post-dose on Day -1
  * hours 0 (pre-dose) 1, 2, 4, 6, 8, 12, 20, 24, 25, 26, 28, 30, 32, 36, 44, 48, 144, 192, 240, 312, 384, 456, 528, 600, 672 post injections 1 and 4
  * hours 0 (pre-dose) 1, 2, 4, 6, 8, 12, 20, 24, 25, 26, 28, 30, 32, 36, 44, 48, 144, 192, 240, 312, 384, 456, 528, 600, 672, 846, 1008, 1200, 1344 post injection 6
Time Frame: Day -1, Days 1-29, 85-113, 141-197
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Group 1 (8 mg) RBP-6000: 50 mg | Group 2 (12 mg) RBP-6000: 100 mg | Group 3 (24 mg) RBP-6000: 200 mg | Group 4 (8 mg) RBP-6000: 100 mg | Group 5 (14 mg) RBP-6000: 200 mg | Group 6 (8-24 mg) RBP-6000: 300 mg
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 14
hr*ng/mL
  Sublingual Period (0-24 hours) | 28.452 (7.9415) | 40.971 (12.6823) | 63.019 (16.4068) | 30.029 (12.8676) | 46.681 (11.8403) | 46.628 (23.2554)
  Initial Burst: Injection 1 (0-48 hours) | 46.855 (11.5533) | 72.453 (25.4451) | 109.029 (30.2598) | 62.395 (20.3054) | 104.868 (22.6943) | 164.511 (47.8237)
  Initial Burst: Injection 4 (0-48 hours): number analyzed (Participants) | 11 | 11 | 11 | 10 | 11 | 6
  Initial Burst: Injection 4 (0-48 hours) | 69.845 (24.4947) | 113.347 (29.7760) | 185.535 (48.2330) | 98.566 (17.8092) | 172.421 (29.3259) | 381.729 (81.4365)
  Initial Burst: Injection 6 (0-48 hours): number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1
  Initial Burst: Injection 6 (0-48 hours) |  |  |  |  | 216.540 (48.7904) | 320.159
  Plateau: Injection 1 (2-28 days): number analyzed (Participants) | 11 | 14 | 14 | 9 | 13 | 10
  Plateau: Injection 1 (2-28 days) | 208.013 (43.2691) | 395.450 (115.3659) | 541.226 (193.6220) | 368.925 (137.2231) | 648.344 (217.2051) | 926.110 (285.6452)
  Plateau: Injection 4 (2-28 days): number analyzed (Participants) | 10 | 12 | 10 | 9 | 10 | 5
  Plateau: Injection 4 (2-28 days) | 596.568 (227.2414) | 1142.046 (380.1915) | 1807.403 (441.0377) | 1073.201 (240.7532) | 1859.204 (477.7799) | 3426.313 (672.5864)
  Plateau: Injection 6 (2-28 days): number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1
  Plateau: Injection 6 (2-28 days) |  |  |  |  | 2209.11 | 3460.459
  Overall: Injection 1 (0-24 hours): number analyzed (Participants) | 15 | 15 | 14 | 15 | 12 | 14
  Overall: Injection 1 (0-24 hours) | 24.922 (6.4450) | 36.981 (14.3565) | 55.291 (17.0179) | 31.747 (13.2180) | 50.034 (11.4899) | 85.090 (28.7163)
  Overall: Injection 1 (0-28 days): number analyzed (Participants) | 15 | 14 | 13 | 14 | 14 | 11
  Overall: Injection 1 (0-28 days) | 246.650 (54.9881) | 461.366 (142.2166) | 642.010 (228.0284) | 413.438 (133.0365) | 756.053 (233.8099) | 1268.012 (389.6719)
  Overall: Injection 4 (0-24 hours): number analyzed (Participants) | 11 | 12 | 11 | 10 | 8 | 7
  Overall: Injection 4 (0-24 hours) | 35.250 (14.5405) | 56.231 (15.6411) | 91.197 (27.4005) | 47.633 (9.6147) | 81.417 (18.3829) | 178.109 (43.2176)
  Overall: Injection 4 (0-28 days): number analyzed (Participants) | 10 | 11 | 9 | 8 | 7 | 2
  Overall: Injection 4 (0-28 days) | 667.611 (254.2712) | 1272.047 (434.1013) | 1932.068 (455.1540) | 1275.098 (252.8500) | 2051.989 (466.6935) | 3230.873 (430.6718)
  Overall: Injection 6 (0-24 hours): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Overall: Injection 6 (0-24 hours) |  |  |  |  |  | 155.779
  Overall: Injection 6 (0-28 days): number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0
  Overall: Injection 6 (0-28 days) |  |  |  |  | 2585.976 (276.6695) |

4. Primary Outcome: Buprenorphine PK: Average Plasma Concentration (Cavg)
Description: Cavg was defined as the AUC (timeframe)/timeframe. For example, the sublingual steady-state Cavg reading on Day -1 = AUC0-24/ 24 hours
  Results are reported across three timeframes:
  * Sublingual Period (Day -1 dose of SUBUTEX): a steady-state reading.
  * Plateau Parameters (Days 3-29 relative to RBP-6000 injections 1, 4 and 6)
  * Overall Parameters (Days 1-29 relative to RBP-6000 injections 1, 4 and 6)
  The PK sampling schedule was
  * hour 0 (predose) on days -7 to -1,
  * hours 0.5, 1,2,4,6, 8,12, 24 post-dose on Day -1
  * hours 0 (pre-dose) 1, 2, 4, 6, 8, 12, 20, 24, 25, 26, 28, 30, 32, 36, 44, 48, 144, 192, 240, 312, 384, 456, 528, 600, 672 post injections 1 and 4
  * hours 0 (pre-dose) 1, 2, 4, 6, 8, 12, 20, 24, 25, 26, 28, 30, 32, 36, 44, 48, 144, 192, 240, 312, 384, 456, 528, 600, 672, 846, 1008, 1200, 1344 post injection 6
Time Frame: Day -1, Days 1-29, 85-113, 141-197
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1 (8 mg) RBP-6000: 50 mg | Group 2 (12 mg) RBP-6000: 100 mg | Group 3 (24 mg) RBP-6000: 200 mg | Group 4 (8 mg) RBP-6000: 100 mg | Group 5 (14 mg) RBP-6000: 200 mg | Group 6 (8-24 mg) RBP-6000: 300 mg
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 14
ng/mL
  Sublingual Period | 1.186 (0.3309) | 1.707 (0.5284) | 2.626 (0.6836) | 1.251 (0.5362) | 1.945 (0.4933) | 1.943 (0.9690)
  Plateau: Injection 1: number analyzed (Participants) | 11 | 14 | 14 | 9 | 13 | 10
  Plateau: Injection 1 | 0.333 (0.0693) | 0.634 (0.1849) | 0.867 (0.3103) | 0.591 (0.2199) | 1.039 (0.3481) | 1.484 (0.4578)
  Plateau: Injection 4: number analyzed (Participants) | 10 | 12 | 10 | 9 | 10 | 5
  Plateau: Injection 4 | 0.954 (0.3642) | 1.830 (0.6093) | 2.896 (0.7068) | 1.720 (0.3858) | 2.979 (0.7657) | 5.491 (1.0779)
  Plateau: Injection 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1
  Plateau: Injection 6 |  |  |  |  | 3.540 | 5.546
  Overall: Injection 1: number analyzed (Participants) | 15 | 14 | 13 | 14 | 14 | 11
  Overall: Injection 1 | 0.367 (0.0818) | 0.687 (0.2116) | 0.955 (0.3393) | 0.615 (0.1980) | 1.125 (0.3331) | 1.887 (0.5799)
  Overall: Injection 4: number analyzed (Participants) | 10 | 11 | 9 | 8 | 7 | 2
  Overall: Injection 4 | 0.993 (0.3784) | 1.893 (0.6460) | 2.875 (0.6773) | 1.897 (0.3763) | 3.054 (0.6945) | 4.808 (0.6409)
  Overall: Injection 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0
  Overall: Injection 6 |  |  |  |  | 3.848 (0.4117) |

5. Primary Outcome: Buprenorphine PK: Maximum Observed Plasma Concentration (Cmax)
Description: Maximum observed plasma concentration, determined directly from individual concentration time data.
  Results are reported across four timeframes:
  * Sublingual Period (Day -1 dose of SUBUTEX): a steady-state reading at hours 0-24.
  * Initial Burst Parameters (Days 1-2 relative to RBP-6000 injections 1, 4 and 6) at hours 0-48
  * Plateau Parameters (Days 3-29 relative to RBP-6000 injections 1, 4 and 6) at hours 48-672
  * Overall Parameters (Days 1-29 relative to RBP-6000 injections 1, 4 and 6)
  The PK sampling schedule was
  * hour 0 (predose) on days -7 to -1,
  * hours 0.5, 1,2,4,6, 8,12, 24 post-dose on Day -1
  * hours 0 (pre-dose) 1, 2, 4, 6, 8, 12, 20, 24, 25, 26, 28, 30, 32, 36, 44, 48, 144, 192, 240, 312, 384, 456, 528, 600, 672 post injections 1 and 4
  * hours 0 (pre-dose) 1, 2, 4, 6, 8, 12, 20, 24, 25, 26, 28, 30, 32, 36, 44, 48, 144, 192, 240, 312, 384, 456, 528, 600, 672, 846, 1008, 1200, 1344 post injection 6
Time Frame: Day -1, Days 1-29, 85-113, 141-197
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1 (8 mg) RBP-6000: 50 mg | Group 2 (12 mg) RBP-6000: 100 mg | Group 3 (24 mg) RBP-6000: 200 mg | Group 4 (8 mg) RBP-6000: 100 mg | Group 5 (14 mg) RBP-6000: 200 mg | Group 6 (8-24 mg) RBP-6000: 300 mg
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 14
ng/mL
  Sublingual Period (0-24 hours) | 3.521 (1.0407) | 5.350 (1.7340) | 7.571 (3.0928) | 3.964 (1.9131) | 5.260 (1.5595) | 5.813 (3.4264)
  Initial Burst: Injection 1 (0-48 hours) | 1.352 (0.4641) | 1.916 (0.6773) | 2.755 (0.7630) | 1.686 (0.6200) | 2.861 (0.7136) | 4.817 (1.4337)
  Initial Burst: Injection 4 (0-48 hours): number analyzed (Participants) | 11 | 12 | 11 | 10 | 11 | 7
  Initial Burst: Injection 4 (0-48 hours) | 2.085 (1.4381) | 2.958 (0.9624) | 4.526 (1.3078) | 2.549 (0.4797) | 4.404 (0.9231) | 9.637 (2.3409)
  Initial Burst: Injection 6 (0-48 hours): number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1
  Initial Burst: Injection 6 (0-48 hours) |  |  |  |  | 5.015 (0.8980) | 7.140
  Plateau: Injection 1 (2-28 days): number analyzed (Participants) | 15 | 15 | 14 | 14 | 15 | 13
  Plateau: Injection 1 (2-28 days) | 0.853 (0.2687) | 1.518 (0.8167) | 2.018 (0.6205) | 1.174 (0.3432) | 2.112 (0.6935) | 2.975 (0.8839)
  Plateau: Injection 4 (2-28 days): number analyzed (Participants) | 11 | 12 | 11 | 10 | 11 | 6
  Plateau: Injection 4 (2-28 days) | 1.384 (0.4767) | 2.590 (0.8536) | 3.776 (0.8970) | 2.211 (0.3824) | 3.780 (0.6646) | 7.452 (1.6913)
  Plateau: Injection 6 (2-28 days): number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1
  Plateau: Injection 6 (2-28 days) |  |  |  |  | 4.650 (0.8910) | 6.550
  Overall: Injection 1: number analyzed (Participants) | 15 | 15 | 14 | 15 | 15 | 14
  Overall: Injection 1 | 1.352 (0.4641) | 2.023 (0.8251) | 2.732 (0.7866) | 1.686 (0.6200) | 2.861 (0.7136) | 4.817 (1.4337)
  Overall: Injection 4: number analyzed (Participants) | 11 | 12 | 11 | 10 | 11 | 7
  Overall: Injection 4 | 2.085 (1.4381) | 3.066 (0.8658) | 4.526 (1.3078) | 2.554 (0.4775) | 4.404 (0.9231) | 9.637 (2.3409)
  Overall: Injection 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1
  Overall: Injection 6 |  |  |  |  | 5.015 (0.8980) | 7.140

6. Primary Outcome: Buprenorphine PK: Minimum Observed Plasma Concentration (Cmin)
Description: Minimum observed plasma concentration, determined directly from individual concentration time data.
  Results are reported across three timeframes:
  * Sublingual Period (Day -1 dose of SUBUTEX): a steady-state reading at hours 0-24.
  * Plateau Parameters (Days 3-29 relative to RBP-6000 injections 1, 4 and 6) at hours 48-672
  * Overall Parameters (Days 1-29 relative to RBP-6000 injections 1, 4 and 6)
  The PK sampling schedule was
  * hour 0 (predose) on days -7 to -1,
  * hours 0.5, 1,2,4,6, 8,12, 24 post-dose on Day -1
  * hours 0 (pre-dose) 1, 2, 4, 6, 8, 12, 20, 24, 25, 26, 28, 30, 32, 36, 44, 48, 144, 192, 240, 312, 384, 456, 528, 600, 672 post injections 1 and 4
  * hours 0 (pre-dose) 1, 2, 4, 6, 8, 12, 20, 24, 25, 26, 28, 30, 32, 36, 44, 48, 144, 192, 240, 312, 384, 456, 528, 600, 672, 846, 1008, 1200, 1344 post injection 6
Time Frame: Day -1, Days 1-29, 85-113, 141-197
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1 (8 mg) RBP-6000: 50 mg | Group 2 (12 mg) RBP-6000: 100 mg | Group 3 (24 mg) RBP-6000: 200 mg | Group 4 (8 mg) RBP-6000: 100 mg | Group 5 (14 mg) RBP-6000: 200 mg | Group 6 (8-24 mg) RBP-6000: 300 mg
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 14
ng/mL
  Sublingual Period (0-24 hours) | 0.524 (0.2212) | 0.806 (0.3638) | 1.385 (0.4806) | 0.568 (0.2367) | 0.920 (0.2800) | 0.927 (0.4667)
  Plateau: Injection 1 (2-28 days): number analyzed (Participants) | 15 | 15 | 14 | 14 | 15 | 13
  Plateau: Injection 1 (2-28 days) | 0.206 (0.0556) | 0.388 (0.1145) | 0.600 (0.2623) | 0.388 (0.1554) | 0.714 (0.2315) | 1.244 (0.4455)
  Plateau: Injection 4 (2-28 days): number analyzed (Participants) | 11 | 12 | 11 | 10 | 11 | 6
  Plateau: Injection 4 (2-28 days) | 0.791 (0.3017) | 1.434 (0.3706) | 2.575 (0.6439) | 1.552 (0.3448) | 2.498 (0.7269) | 4.600 (0.7743)
  Plateau: Injection 6 (2-28 days): number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1
  Plateau: Injection 6 (2-28 days) |  |  |  |  | 3.325 (0.1485) | 4.810
  Overall: Injection 1: number analyzed (Participants) | 15 | 15 | 14 | 15 | 15 | 14
  Overall: Injection 1 | 0.206 (0.0556) | 0.375 (0.1001) | 0.589 (0.2522) | 0.410 (0.1955) | 0.700 (0.2196) | 0.836 (0.3756)
  Overall: Injection 4: number analyzed (Participants) | 11 | 12 | 11 | 10 | 11 | 7
  Overall: Injection 4 | 0.557 (0.1559) | 1.263 (0.3574) | 2.121 (0.4689) | 1.180 (0.2803) | 2.256 (0.6472) | 4.043 (0.6936)
  Overall: Injection 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1
  Overall: Injection 6 |  |  |  |  | 2.910 (0.7354) | 4.290

7. Primary Outcome: Buprenorphine PK: Swing of Plasma Concentrations
Description: The swing of buprenorphine plasma concentrations calculated as (Cmax-Cmin)/Cmin within the dosing interval.
  Cmax=maximum plasma concentration Cmin=minimum plasma concentration
  Results are reported across three timeframes:
  * Sublingual Period (Day -1 dose of SUBUTEX): a steady-state reading.
  * Plateau Parameters (Days 3-29 relative to RBP-6000 injections 1, 4 and 6)
  * Overall Parameters (Days 1-29 relative to RBP-6000 injections 1, 4 and 6)
  The PK sampling schedule was
  * hour 0 (predose) on days -7 to -1,
  * hours 0.5, 1,2,4,6, 8,12, 24 post-dose on Day -1
  * hours 0 (pre-dose) 1, 2, 4, 6, 8, 12, 20, 24, 25, 26, 28, 30, 32, 36, 44, 48, 144, 192, 240, 312, 384, 456, 528, 600, 672 post injections 1 and 4
  * hours 0 (pre-dose) 1, 2, 4, 6, 8, 12, 20, 24, 25, 26, 28, 30, 32, 36, 44, 48, 144, 192, 240, 312, 384, 456, 528, 600, 672, 846, 1008, 1200, 1344 post injection 6
Time Frame: Day -1, Days 1-29, 85-113, 141-197
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of Cmin
Arm/Group | Group 1 (8 mg) RBP-6000: 50 mg | Group 2 (12 mg) RBP-6000: 100 mg | Group 3 (24 mg) RBP-6000: 200 mg | Group 4 (8 mg) RBP-6000: 100 mg | Group 5 (14 mg) RBP-6000: 200 mg | Group 6 (8-24 mg) RBP-6000: 300 mg
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 14
percentage of Cmin
  Sublingual Period | 656.884 (303.7135) | 665.742 (314.6530) | 493.475 (273.1229) | 597.543 (136.8431) | 500.322 (183.7474) | 534.280 (217.8816)
  Plateau: Injection 1: number analyzed (Participants) | 15 | 15 | 14 | 14 | 15 | 13
  Plateau: Injection 1 | 332.132 (127.9638) | 295.987 (229.0036) | 253.417 (61.2944) | 223.388 (94.3116) | 197.895 (49.3822) | 147.463 (66.0341)
  Plateau: Injection 4: number analyzed (Participants) | 11 | 12 | 11 | 10 | 11 | 6
  Plateau: Injection 4 | 79.731 (27.3175) | 84.772 (48.3724) | 47.479 (10.5422) | 44.874 (18.5656) | 57.889 (30.3975) | 61.481 (24.0339)
  Plateau: Injection 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1
  Plateau: Injection 6 |  |  |  |  | 39.390 (20.5703) | 36.175
  Overall: Injection 1: number analyzed (Participants) | 15 | 15 | 14 | 15 | 15 | 14
  Overall: Injection 1 | 586.788 (219.9900) | 440.102 (200.5223) | 399.355 (140.2055) | 350.591 (158.0245) | 336.666 (149.7124) | 548.179 (272.0431)
  Overall: Injection 4: number analyzed (Participants) | 11 | 12 | 11 | 10 | 11 | 7
  Overall: Injection 4 | 279.713 (214.1821) | 147.264 (48.3533) | 112.812 (32.8955) | 120.236 (28.1402) | 103.271 (43.4914) | 138.783 (47.6186)
  Overall: Injection 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1
  Overall: Injection 6 |  |  |  |  | 73.993 (13.1102) | 66.434

8. Primary Outcome: Buprenorphine PK: Time to Maximum Buprenorphine Plasma Concentration (Tmax)
Description: Results are reported across four timeframes:
  * Sublingual Period (Day -1 dose of SUBUTEX): a steady-state reading at hours 0-24.
  * Initial Burst Parameters (Days 1-2 relative to RBP-6000 injections 1, 4 and 6) at hours 0-48
  * Plateau Parameters (Days 3-29 relative to RBP-6000 injections 1, 4 and 6) at hours 48-672
  * Overall Parameters (Days 1-29 relative to RBP-6000 injections 1, 4 and 6) at hours 0-24, hours 0-672
  The PK sampling schedule was
  * hour 0 (predose) on days -7 to -1,
  * hours 0.5, 1,2,4,6, 8,12, 24 post-dose on Day -1
  * hours 0 (pre-dose) 1, 2, 4, 6, 8, 12, 20, 24, 25, 26, 28, 30, 32, 36, 44, 48, 144, 192, 240, 312, 384, 456, 528, 600, 672 post injections 1 and 4
  * hours 0 (pre-dose) 1, 2, 4, 6, 8, 12, 20, 24, 25, 26, 28, 30, 32, 36, 44, 48, 144, 192, 240, 312, 384, 456, 528, 600, 672, 846, 1008, 1200, 1344 post injection 6
Time Frame: Day -1, Days 1-29, 85-113, 141-197
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Group 1 (8 mg) RBP-6000: 50 mg | Group 2 (12 mg) RBP-6000: 100 mg | Group 3 (24 mg) RBP-6000: 200 mg | Group 4 (8 mg) RBP-6000: 100 mg | Group 5 (14 mg) RBP-6000: 200 mg | Group 6 (8-24 mg) RBP-6000: 300 mg
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 14
hours
  Sublingual Period (0-24 hours) | 2.000 [1.00 to 4.00] | 1.017 [0.50 to 2.00] | 1.117 [0.50 to 2.00] | 2.000 [1.00 to 2.00] | 2.000 [0.50 to 2.13] | 2.000 [1.00 to 2.00]
  Initial Burst: Injection 1 (0-48 hours) | 20.000 [4.00 to 20.05] | 20.000 [4.00 to 48.00] | 20.000 [6.00 to 48.00] | 20.000 [4.00 to 48.00] | 20.000 [6.00 to 48.00] | 20.000 [4.00 to 32.00]
  Initial Burst: Injection 4 (0-48 hours): number analyzed (Participants) | 11 | 11 | 11 | 10 | 11 | 7
  Initial Burst: Injection 4 (0-48 hours) | 20.000 [2.00 to 24.00] | 20.000 [4.00 to 30.07] | 20.083 [8.00 to 30.08] | 24.000 [4.00 to 48.03] | 24.000 [4.00 to 48.00] | 24.000 [4.00 to 36.00]
  Initial Burst: Injection 6 (0-48 hours): number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1
  Initial Burst: Injection 6 (0-48 hours) |  |  |  |  | 24.000 [24.00 to 24.00] | 24.350 [24.35 to 24.35]
  Plateau: Injection 1 (2-28 days): number analyzed (Participants) | 15 | 15 | 14 | 14 | 15 | 13
  Plateau: Injection 1 (2-28 days) | 48.000 [48.00 to 48.00] | 48.000 [48.00 to 457.15] | 48.000 [48.00 to 49.10] | 48.000 [48.00 to 48.07] | 48.000 [48.00 to 48.07] | 48.000 [48.00 to 532.55]
  Plateau: Injection 4 (2-28 days): number analyzed (Participants) | 11 | 12 | 11 | 10 | 11 | 6
  Plateau: Injection 4 (2-28 days) | 48.000 [48.00 to 48.07] | 48.000 [48.00 to 315.95] | 48.000 [48.00 to 49.12] | 48.000 [48.00 to 629.07] | 48.000 [48.00 to 485.17] | 48.000 [48.00 to 436.75]
  Plateau: Injection 6 (2-28 days): number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1
  Plateau: Injection 6 (2-28 days) |  |  |  |  | 48.000 [48.00 to 48.00] | 48.000 [48.00 to 48.00]
  Overall: Injection 1 (0-28 days): number analyzed (Participants) | 15 | 15 | 14 | 15 | 15 | 14
  Overall: Injection 1 (0-28 days) | 20.000 [4.00 to 20.05] | 20.000 [4.00 to 414.17] | 20.000 [6.00 to 30.00] | 20.000 [4.00 to 48.00] | 20.000 [6.00 to 48.00] | 20.000 [4.00 to 32.00]
  Overall: Injection 4 (0-28 days): number analyzed (Participants) | 11 | 12 | 11 | 10 | 11 | 7
  Overall: Injection 4 (0-28 days) | 20.000 [2.00 to 24.00] | 20.000 [12.00 to 315.95] | 20.083 [8.00 to 30.08] | 24.000 [4.00 to 529.83] | 24.000 [4.00 to 48.00] | 24.000 [4.00 to 36.00]
  Overall: Injection 6 (0-28 days): number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1
  Overall: Injection 6 (0-28 days) |  |  |  |  | 24.000 [24.00 to 24.00] | 24.350 [24.35 to 24.35]

9. Primary Outcome: Buprenorphine PK: Accumulation Index in Terms of Area Under the Curve (Rac(AUC))
Description: Accumulation index in terms of AUC calculated as ratio of AUCtau Injection 4/ AUCtau Injection 1. AUCtau = area under plasma concentration time curve over the dosing interval tau (for SC RBP-6000, tau=28 days).
Time Frame: Days 1-28, 85-113
Population: PK population of participants with data at both timepoints
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Group 1 (8 mg) RBP-6000: 50 mg | Group 2 (12 mg) RBP-6000: 100 mg | Group 3 (24 mg) RBP-6000: 200 mg | Group 4 (8 mg) RBP-6000: 100 mg | Group 5 (14 mg) RBP-6000: 200 mg | Group 6 (8-24 mg) RBP-6000: 300 mg
Number analyzed (Participants) | 10 | 11 | 9 | 8 | 7 | 2
ratio | 2.580 (0.9662) | 2.738 (0.5104) | 3.456 (0.9296) | 3.379 (0.9182) | 2.837 (0.8660) | 3.573 (0.5660)

10. Primary Outcome: Buprenorphine PK: Accumulation Index in Terms of Maximum Observed Plasma Drug Concentration (Rac(Cmax))
Description: Accumulation index in terms of Cmax calculated as ratio of Cmax Injection 4/ Cmax Injection 1.
Time Frame: Days 1-28, 85-113
Population: PK population of participants with data at both timepoints
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Group 1 (8 mg) RBP-6000: 50 mg | Group 2 (12 mg) RBP-6000: 100 mg | Group 3 (24 mg) RBP-6000: 200 mg | Group 4 (8 mg) RBP-6000: 100 mg | Group 5 (14 mg) RBP-6000: 200 mg | Group 6 (8-24 mg) RBP-6000: 300 mg
Number analyzed (Participants) | 11 | 12 | 11 | 10 | 11 | 7
ratio | 1.380 (0.4610) | 1.560 (0.5322) | 1.766 (0.5407) | 1.729 (0.6106) | 1.559 (0.2642) | 1.908 (0.4411)

11. Primary Outcome: Buprenorphine PK: Apparent Clearance at Steady-State (CLss/F) Following Injections 4 and 6
Description: Apparent clearance at steady-state (CLss/F) = Dose / AUCtau (tau was 28 days).
Time Frame: Days 85-113, 141-169
Population: PK population
Measure: Mean (Standard Deviation); unit: L/hour
Arm/Group | Group 1 (8 mg) RBP-6000: 50 mg | Group 2 (12 mg) RBP-6000: 100 mg | Group 3 (24 mg) RBP-6000: 200 mg | Group 4 (8 mg) RBP-6000: 100 mg | Group 5 (14 mg) RBP-6000: 200 mg | Group 6 (8-24 mg) RBP-6000: 300 mg
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 14
L/hour
  Injection 4: number analyzed (Participants) | 11 | 12 | 11 | 10 | 8 | 5
  Injection 4 | 85.543 (34.6133) | 85.043 (21.9189) | 105.155 (23.4377) | 87.404 (21.0436) | 105.390 (29.3714) | 80.860 (15.8555)
  Injection 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1
  Injection 6 |  |  |  |  | 77.749 (8.3342) | 79.777

12. Primary Outcome: Buprenorphine PK: Area Under Plasma Concentration Time Curve From Time Zero Of Injection 4 (AUC0-∞)
Description: Area under plasma concentration time curve from time zero of Injection 4 extrapolated to infinity; calculated for Injection 4 (last injection) in subjects not participating in PET imaging sub-study only as:
  (AUC0-∞ was reported if the coefficient of determination R2 was at least 0.8 and the extrapolated area is less than 25%). A minimum of 5 data points was required. AUC up to the last measurable concentration (AUClast) was calculated by using the linear trapezoidal rule.
Time Frame: Days 85-113
Population: PK population of participants whose data met requirements.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Group 1 (8 mg) RBP-6000: 50 mg | Group 2 (12 mg) RBP-6000: 100 mg | Group 3 (24 mg) RBP-6000: 200 mg | Group 4 (8 mg) RBP-6000: 100 mg | Group 5 (14 mg) RBP-6000: 200 mg | Group 6 (8-24 mg) RBP-6000: 300 mg
Number analyzed (Participants) | 2 | 1 | 0 | 0 | 0 | 0
hr*ng/mL | 2280.295 (17.4444) | 3521.376 |  |  |  |

13. Primary Outcome: Buprenorphine PK: Terminal Phase Half Life (t1/2) Calculated For Injection 4
Description: The terminal phase half life calculated for Injection 4 in subjects not participating in PET imaging sub-study. The t1/2 was reported only if the coefficient of determination R2 was at least 0.8.
Time Frame: Days 85-113
Population: PK population of participants whose data met requirements.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Group 1 (8 mg) RBP-6000: 50 mg | Group 2 (12 mg) RBP-6000: 100 mg | Group 3 (24 mg) RBP-6000: 200 mg | Group 4 (8 mg) RBP-6000: 100 mg | Group 5 (14 mg) RBP-6000: 200 mg | Group 6 (8-24 mg) RBP-6000: 300 mg
Number analyzed (Participants) | 2 | 1 | 0 | 0 | 0 | 0
hours | 550.329 (36.7325) | 138.238 |  |  |  |

14. Primary Outcome: Norbuprenorphine PK: % Fluctuation
Description: % Fluctuation was defined as the degree of fluctuation of norbuprenorphine plasma concentrations calculated as (Cmax-Cmin)/Cavg*100, expressed as a percentage. Cmax=maximum plasma concentration Cmin=minimum plasma concentration Cavg = average plasma concentration
  Results are reported across three timeframes:
  * Sublingual Period (Day -1 dose of SUBUTEX): a steady-state reading.
  * Plateau Parameters (Days 3-29 relative to RBP-6000 injections 1, 4 and 6)
  * Overall Parameters (Days 1-29 relative to RBP-6000 injections 1, 4 and 6)
  The PK sampling schedule was
  * hour 0 (predose) on days -7 to -1,
  * hours 0.5, 1,2,4,6, 8,12, 24 post-dose on Day -1
  * hours 0 (pre-dose) 1, 2, 4, 6, 8, 12, 20, 24, 25, 26, 28, 30, 32, 36, 44, 48, 144, 192, 240, 312, 384, 456, 528, 600, 672 post injections 1 and 4
  * hours 0 (pre-dose) 1, 2, 4, 6, 8, 12, 20, 24, 25, 26, 28, 30, 32, 36, 44, 48, 144, 192, 240, 312, 384, 456, 528, 600, 672, 846, 1008, 1200, 1344 post injection 6
Time Frame: Day -1, Days 1-29, 85-113, 141-197
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: % of average concentration
Arm/Group | Group 1 (8 mg) RBP-6000: 50 mg | Group 2 (12 mg) RBP-6000: 100 mg | Group 3 (24 mg) RBP-6000: 200 mg | Group 4 (8 mg) RBP-6000: 100 mg | Group 5 (14 mg) RBP-6000: 200 mg | Group 6 (8-24 mg) RBP-6000: 300 mg
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 14
% of average concentration
  Sublingual Period: number analyzed (Participants) | 15 | 15 | 12 | 13 | 10 | 14
  Sublingual Period | 69.798 (21.5137) | 94.132 (43.7842) | 79.225 (19.2173) | 82.834 (29.0182) | 89.832 (31.3881) | 71.213 (18.7721)
  Plateau: Injection 1: number analyzed (Participants) | 14 | 14 | 13 | 13 | 15 | 12
  Plateau: Injection 1 | 577.952 (119.5038) | 475.800 (149.9103) | 504.540 (170.1714) | 403.009 (115.9346) | 407.217 (160.6071) | 354.764 (136.5715)
  Plateau: Injection 4: number analyzed (Participants) | 10 | 11 | 9 | 7 | 8 | 5
  Plateau: Injection 4 | 114.801 (33.7254) | 127.106 (64.0505) | 110.567 (42.0264) | 77.455 (24.7664) | 101.898 (28.8808) | 83.579 (18.6265)
  Plateau: Injection 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1
  Plateau: Injection 6 |  |  |  |  | 91.763 | 242.246
  Overall: Injection 1: number analyzed (Participants) | 11 | 12 | 13 | 14 | 14 | 11
  Overall: Injection 1 | 612.998 (141.7474) | 502.856 (101.2508) | 685.962 (195.9687) | 497.361 (138.6539) | 609.481 (145.8650) | 468.074 (186.0526)
  Overall: Injection 4: number analyzed (Participants) | 10 | 11 | 9 | 8 | 7 | 2
  Overall: Injection 4 | 128.273 (31.6391) | 131.080 (57.4294) | 127.005 (37.8487) | 95.960 (18.6296) | 131.650 (43.6260) | 102.192 (12.2405)
  Overall: Injection 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0
  Overall: Injection 6 |  |  |  |  | 94.048 (7.4553) |

15. Primary Outcome: Norbuprenorphine PK: Area Under Plasma Concentration Time Curves (AUC)
Description: as for outcome 3
Time Frame: Day -1, Days 1-29, 85-113, 141-197
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Group 1 (8 mg) RBP-6000: 50 mg | Group 2 (12 mg) RBP-6000: 100 mg | Group 3 (24 mg) RBP-6000: 200 mg | Group 4 (8 mg) RBP-6000: 100 mg | Group 5 (14 mg) RBP-6000: 200 mg | Group 6 (8-24 mg) RBP-6000: 300 mg
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 14
hr*ng/mL
  Sublingual Period (0-24 hours): number analyzed (Participants) | 15 | 15 | 12 | 13 | 10 | 14
  Sublingual Period (0-24 hours) | 42.536 (17.9975) | 72.339 (35.1371) | 134.739 (40.4214) | 49.312 (22.6050) | 65.558 (25.0632) | 98.407 (81.7085)
  Initial Burst: Injection 1 (0-48 hours) | 60.834 (27.8301) | 98.705 (54.0709) | 180.685 (53.1546) | 69.878 (26.1289) | 131.277 (82.0351) | 148.016 (97.0872)
  Initial Burst: Injection 4 (0-48 hours): number analyzed (Participants) | 11 | 11 | 11 | 10 | 11 | 6
  Initial Burst: Injection 4 (0-48 hours) | 15.435 (8.0734) | 29.401 (16.3007) | 50.185 (19.6558) | 30.755 (11.0344) | 45.941 (24.8979) | 101.888 (39.8768)
  Initial Burst: Injection 6 (0-48 hours): number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1
  Initial Burst: Injection 6 (0-48 hours) |  |  |  |  | 59.352 (2.2741) | 90.719
  Plateau: Injection 1 (2-28 days): number analyzed (Participants) | 14 | 14 | 13 | 13 | 15 | 12
  Plateau: Injection 1 (2-28 days) | 122.265 (43.4215) | 209.679 (85.5994) | 384.101 (133.4394) | 197.483 (59.5501) | 295.342 (142.3582) | 513.577 (322.8520)
  Plateau: Injection 4 (2-28 days): number analyzed (Participants) | 10 | 11 | 9 | 7 | 8 | 5
  Plateau: Injection 4 (2-28 days) | 166.360 (82.1264) | 523.076 (431.7284) | 519.103 (236.8835) | 410.621 (146.1564) | 550.225 (215.6699) | 1208.505 (463.9637)
  Plateau: Injection 6 (2-28 days): number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1
  Plateau: Injection 6 (2-28 days) |  |  |  |  | 537.212 | 592.199
  Overall: Injection 1 (0-24 hours): number analyzed (Participants) | 15 | 15 | 14 | 15 | 12 | 14
  Overall: Injection 1 (0-24 hours) | 32.465 (14.2953) | 52.878 (28.0773) | 99.040 (30.8899) | 37.446 (15.9959) | 68.660 (38.8033) | 80.525 (51.3662)
  Overall: Injection 1 (0-28 days): number analyzed (Participants) | 11 | 12 | 13 | 14 | 14 | 11
  Overall: Injection 1 (0-28 days) | 181.912 (81.6100) | 343.357 (150.5029) | 541.539 (176.5176) | 261.745 (81.3672) | 426.283 (224.4167) | 688.487 (429.8748)
  Overall: Injection 4 (0-24 hours): number analyzed (Participants) | 11 | 12 | 11 | 10 | 8 | 7
  Overall: Injection 4 (0-24 hours) | 6.274 (2.7973) | 15.199 (11.7793) | 22.870 (9.3521) | 13.807 (5.3021) | 16.301 (6.4778) | 43.722 (16.4542)
  Overall: Injection 4 (0-28 days): number analyzed (Participants) | 10 | 11 | 9 | 8 | 7 | 2
  Overall: Injection 4 (0-28 days) | 182.405 (91.5308) | 557.707 (471.2095) | 570.958 (254.4439) | 452.892 (152.6941) | 673.245 (167.1460) | 658.609 (159.7954)
  Overall: Injection 6 (0-24 hours): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Overall: Injection 6 (0-24 hours) |  |  |  |  |  | 37.093
  Overall: Injection 6 (0-28 days): number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0
  Overall: Injection 6 (0-28 days) |  |  |  |  | 814.570 (306.2799) |

16. Primary Outcome: Norbuprenorphine PK: Average Plasma Concentration (Cavg)
Description: as for outcome 4
Time Frame: Day -1, Days 1-29, 85-113, 141-197
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1 (8 mg) RBP-6000: 50 mg | Group 2 (12 mg) RBP-6000: 100 mg | Group 3 (24 mg) RBP-6000: 200 mg | Group 4 (8 mg) RBP-6000: 100 mg | Group 5 (14 mg) RBP-6000: 200 mg | Group 6 (8-24 mg) RBP-6000: 300 mg
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 14
ng/mL
  Sublingual Period: number analyzed (Participants) | 15 | 15 | 12 | 13 | 10 | 14
  Sublingual Period | 1.772 (0.7499) | 3.014 (1.4640) | 5.614 (1.6842) | 2.055 (0.9419) | 2.732 (1.0443) | 4.100 (3.4045)
  Plateau: Injection 1: number analyzed (Participants) | 14 | 14 | 13 | 13 | 15 | 12
  Plateau: Injection 1 | 0.196 (0.0696) | 0.336 (0.1372) | 0.616 (0.2138) | 0.316 (0.0954) | 0.473 (0.2281) | 0.823 (0.5174)
  Plateau: Injection 4: number analyzed (Participants) | 10 | 11 | 9 | 7 | 8 | 5
  Plateau: Injection 4 | 0.267 (0.1316) | 0.838 (0.6919) | 0.832 (0.3796) | 0.658 (0.2342) | 0.882 (0.3456) | 1.937 (0.7435)
  Plateau: Injection 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1
  Plateau: Injection 6 |  |  |  |  | 0.861 | 0.949
  Overall: Injection 1: number analyzed (Participants) | 11 | 12 | 13 | 14 | 14 | 11
  Overall: Injection 1 | 0.271 (0.1214) | 0.511 (0.2240) | 0.806 (0.2627) | 0.390 (0.1211) | 0.634 (0.3340) | 1.025 (0.6397)
  Overall: Injection 4: number analyzed (Participants) | 10 | 11 | 9 | 8 | 7 | 2
  Overall: Injection 4 | 0.271 (0.1362) | 0.830 (0.7012) | 0.850 (0.3786) | 0.674 (0.2272) | 1.002 (0.2487) | 0.980 (0.2378)
  Overall: Injection 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0
  Overall: Injection 6 |  |  |  |  | 1.212 (0.4558) |

17. Primary Outcome: Norbuprenorphine PK: Maximum Observed Plasma Concentration (Cmax)
Description: as for outcome 5
Time Frame: Day -1, Days 1-29, 85-113, 141-197
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1 (8 mg) RBP-6000: 50 mg | Group 2 (12 mg) RBP-6000: 100 mg | Group 3 (24 mg) RBP-6000: 200 mg | Group 4 (8 mg) RBP-6000: 100 mg | Group 5 (14 mg) RBP-6000: 200 mg | Group 6 (8-24 mg) RBP-6000: 300 mg
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 14
ng/mL
  Sublingual Period (0-24 hours) | 2.559 (1.0590) | 4.941 (2.5414) | 8.515 (2.3854) | 3.268 (1.6946) | 5.268 (1.9934) | 5.820 (4.7007)
  Initial Burst: Injection 1 (0-48 hours) | 1.674 (0.7498) | 2.704 (1.3861) | 5.335 (1.7751) | 1.965 (0.7884) | 3.878 (2.1658) | 4.496 (3.0242)
  Initial Burst: Injection 4 (0-48 hours): number analyzed (Participants) | 11 | 12 | 11 | 10 | 11 | 7
  Initial Burst: Injection 4 (0-48 hours) | 0.462 (0.2894) | 0.966 (0.5829) | 1.343 (0.4299) | 0.799 (0.2673) | 1.305 (0.5998) | 2.769 (1.2538)
  Initial Burst: Injection 6 (0-48 hours): number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1
  Initial Burst: Injection 6 (0-48 hours) |  |  |  |  | 1.885 (0.6152) | 2.620
  Plateau: Injection 1 (2-28 days): number analyzed (Participants) | 15 | 15 | 14 | 14 | 15 | 13
  Plateau: Injection 1 (2-28 days) | 1.165 (0.5506) | 1.904 (1.0984) | 3.201 (1.1802) | 1.320 (0.4278) | 2.203 (1.4464) | 3.212 (2.8810)
  Plateau: Injection 4 (2-28 days): number analyzed (Participants) | 11 | 12 | 11 | 10 | 11 | 6
  Plateau: Injection 4 (2-28 days) | 0.464 (0.2903) | 1.423 (1.1714) | 1.387 (0.4635) | 0.926 (0.3107) | 1.420 (0.7152) | 2.710 (1.1727)
  Plateau: Injection 6 (2-28 days): number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1
  Plateau: Injection 6 (2-28 days) |  |  |  |  | 1.885 (0.6152) | 2.620
  Overall: Injection 1: number analyzed (Participants) | 15 | 15 | 14 | 15 | 15 | 14
  Overall: Injection 1 | 1.698 (0.7748) | 2.753 (1.4051) | 5,572 (1.9291) | 1.977 (0.7880) | 3.989 (2.3167) | 4.555 (3.1010)
  Overall: Injection 4: number analyzed (Participants) | 11 | 12 | 11 | 10 | 11 | 7
  Overall: Injection 4 | 0.474 (0.2849) | 1.431 (1.1652) | 1.456 (0.4572) | 0.929 (0.3058) | 1.539 (0.6406) | 2.769 (1.2538)
  Overall: Injection 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1
  Overall: Injection 6 |  |  |  |  | 1.885 (0.6152) | 2.620

18. Primary Outcome: Norbuprenorphine PK: Minimum Observed Plasma Concentration (Cmin)
Description: as for outcome 6
Time Frame: Day -1, Days 1-29, 85-113, 141-197
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1 (8 mg) RBP-6000: 50 mg | Group 2 (12 mg) RBP-6000: 100 mg | Group 3 (24 mg) RBP-6000: 200 mg | Group 4 (8 mg) RBP-6000: 100 mg | Group 5 (14 mg) RBP-6000: 200 mg | Group 6 (8-24 mg) RBP-6000: 300 mg
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 14
ng/mL
  Sublingual Period (0-24 hours) | 1.361 (0.6010) | 2.342 (1.2494) | 4.287 (1.3351) | 1.582 (0.7554) | 2.482 (1.1788) | 2.923 (2.1949)
  Plateau: Injection 1 (2-28 days): number analyzed (Participants) | 15 | 15 | 14 | 14 | 15 | 13
  Plateau: Injection 1 (2-28 days) | 0.057 (0.0202) | 0.099 (0.0447) | 0.162 (0.0827) | 0.119 (0.0592) | 0.177 (0.0919) | 0.258 (0.1289)
  Plateau: Injection 4 (2-28 days): number analyzed (Participants) | 11 | 12 | 11 | 10 | 11 | 6
  Plateau: Injection 4 (2-28 days) | 0.165 (0.0708) | 0.432 (0.4181) | 0.548 (0.2119) | 0.439 (0.1550) | 0.587 (0.3165) | 1.234 (0.5279)
  Plateau: Injection 6 (2-28 days): number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1
  Plateau: Injection 6 (2-28 days) |  |  |  |  | 0.895 (0.3323) | 0.321
  Overall: Injection 1: number analyzed (Participants) | 15 | 15 | 14 | 15 | 15 | 14
  Overall: Injection 1 | 0.057 (0.0202) | 0.098 (0.0441) | 0.162 (0.0827) | 0.152 (0.1427) | 0.177 (0.0919) | 0.301 (0.2180)
  Overall: Injection 4: number analyzed (Participants) | 11 | 12 | 11 | 10 | 11 | 7
  Overall: Injection 4 | 0.125 (0.0539) | 0.327 (0.2592) | 0.461 (0.2292) | 0.349 (0.1609) | 0.459 (0.2191) | 0.982 (0.3281)
  Overall: Injection 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1
  Overall: Injection 6 |  |  |  |  | 0.728 (0.0962) | 0.281

19. Primary Outcome: Norbuprenorphine PK: Swing of Plasma Concentrations
Description: The swing of norbuprenorphine plasma concentrations calculated as (Cmax-Cmin)/Cmin within the dosing interval.
  Cmax=maximum plasma concentration Cmin=minimum plasma concentration
  Results are reported across three timeframes:
  * Sublingual Period (Day -1 dose of SUBUTEX): a steady-state reading.
  * Plateau Parameters (Days 3-29 relative to RBP-6000 injections 1, 4 and 6)
  * Overall Parameters (Days 1-29 relative to RBP-6000 injections 1, 4 and 6)
  The PK sampling schedule was
  * hour 0 (predose) on days -7 to -1,
  * hours 0.5, 1,2,4,6, 8,12, 24 post-dose on Day -1
  * hours 0 (pre-dose) 1, 2, 4, 6, 8, 12, 20, 24, 25, 26, 28, 30, 32, 36, 44, 48, 144, 192, 240, 312, 384, 456, 528, 600, 672 post injections 1 and 4
  * hours 0 (pre-dose) 1, 2, 4, 6, 8, 12, 20, 24, 25, 26, 28, 30, 32, 36, 44, 48, 144, 192, 240, 312, 384, 456, 528, 600, 672, 846, 1008, 1200, 1344 post injection 6
Time Frame: Day -1, Days 1-29, 85-113, 141-197
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of Cmin
Arm/Group | Group 1 (8 mg) RBP-6000: 50 mg | Group 2 (12 mg) RBP-6000: 100 mg | Group 3 (24 mg) RBP-6000: 200 mg | Group 4 (8 mg) RBP-6000: 100 mg | Group 5 (14 mg) RBP-6000: 200 mg | Group 6 (8-24 mg) RBP-6000: 300 mg
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 14
percentage of Cmin
  Sublingual Period | 93.472 (33.4835) | 130.823 (74.2916) | 102.059 (29.6116) | 109.416 (42.1913) | 124.601 (45.9786) | 101.558 (38.5511)
  Plateau: Injection 1: number analyzed (Participants) | 15 | 15 | 14 | 14 | 15 | 13
  Plateau: Injection 1 | 1993.328 (1002.6237) | 1871.238 (933.9815) | 2531.386 (1775.8060) | 1188.490 (491.1526) | 1210.967 (874.2858) | 1250.370 (866.1860)
  Plateau: Injection 4: number analyzed (Participants) | 11 | 12 | 11 | 10 | 11 | 6
  Plateau: Injection 4 | 180.340 (82.9960) | 289.316 (271.1318) | 171.673 (98.3404) | 121.682 (62.5967) | 151.990 (82.8360) | 118.215 (42.3788)
  Plateau: Injection 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1
  Plateau: Injection 6 |  |  |  |  | 112.503 (10.1733) | 716.199
  Overall: Injection 1: number analyzed (Participants) | 15 | 15 | 14 | 15 | 15 | 14
  Overall: Injection 1 | 2903.100 (1102.0127) | 2812.484 (1305.9088) | 4477.582 (3470.4282) | 1776.276 (923.9753) | 2355.099 (1345.4616) | 2116.996 (2015.7199)
  Overall: Injection 4: number analyzed (Participants) | 11 | 12 | 11 | 10 | 11 | 7
  Overall: Injection 4 | 322.876 (297.9631) | 379.301 (371.3835) | 265.586 (132.0434) | 186.942 (65.4013) | 272.260 (139.1806) | 173.090 (51.8058)
  Overall: Injection 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1
  Overall: Injection 6 |  |  |  |  | 155.577 (50.7422) | 832.384

20. Primary Outcome: Norbuprenorphine PK: Time to Maximum Buprenorphine Plasma Concentration (Tmax)
Description: as for outcome 8
Time Frame: Day -1, Days 1-29, 85-113, 141-197
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Group 1 (8 mg) RBP-6000: 50 mg | Group 2 (12 mg) RBP-6000: 100 mg | Group 3 (24 mg) RBP-6000: 200 mg | Group 4 (8 mg) RBP-6000: 100 mg | Group 5 (14 mg) RBP-6000: 200 mg | Group 6 (8-24 mg) RBP-6000: 300 mg
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 14
hours
  Sublingual Period (0-24 hours) | 2.000 [0.50 to 4.00] | 1.017 [0.50 to 2.00] | 1.000 [0.50 to 23.58] | 2.000 [0.50 to 12.00] | 2.000 [1.00 to 23.67] | 2.000 [1.00 to 4.00]
  Initial Burst: Injection 1 (0-48 hours) | 8.000 [1.00 to 48.00] | 6.000 [1.00 to 48.00] | 4.000 [1.00 to 30.00] | 12.000 [2.00 to 30.00] | 6.000 [1.00 to 30.00] | 4.000 [1.00 to 36.00]
  Initial Burst: Injection 4 (0-48 hours): number analyzed (Participants) | 11 | 12 | 11 | 10 | 11 | 7
  Initial Burst: Injection 4 (0-48 hours) | 48.000 [1.00 to 48.07] | 48.000 [4.00 to 48.00] | 48.000 [6.00 to 48.10] | 39.000 [8.00 to 48.03] | 24.000 [4.00 to 48.00] | 12.000 [6.00 to 48.00]
  Initial Burst: Injection 6 (0-48 hours): number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1
  Initial Burst: Injection 6 (0-48 hours) |  |  |  |  | 48.000 [48.00 to 48.00] | 48.000 [48.00 to 48.00]
  Plateau: Injection 1 (2-28 days): number analyzed (Participants) | 15 | 15 | 14 | 14 | 15 | 13
  Plateau: Injection 1 (2-28 days) | 48.000 [48.00 to 48.00] | 48.000 [48.00 to 457.15] | 48.000 [48.00 to 48.10] | 48.000 [48.00 to 48.07] | 48.000 [48.00 to 48.07] | 48.000 [48.00 to 48.00]
  Plateau: Injection 4 (2-28 days): number analyzed (Participants) | 11 | 12 | 11 | 10 | 11 | 6
  Plateau: Injection 4 (2-28 days) | 48.000 [48.00 to 408.52] | 96.883 [48.00 to 604.77] | 48.100 [48.00 to 456.80] | 182.808 [48.00 to 629.07] | 167.017 [48.00 to 459.00] | 303.133 [48.00 to 436.75]
  Plateau: Injection 6 (2-28 days): number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1
  Plateau: Injection 6 (2-28 days) |  |  |  |  | 48.000 [48.00 to 48.00] | 48.000 [48.00 to 48.00]
  Overall: Injection 1 (0-28 days): number analyzed (Participants) | 15 | 15 | 14 | 15 | 15 | 14
  Overall: Injection 1 (0-28 days) | 8.000 [0.00 to 48.00] | 6.000 [0.00 to 457.15] | 2.525 [0.00 to 30.00] | 6.000 [0.00 to 30.00] | 4.000 [0.00 to 30.00] | 4.000 [0.00 to 36.00]
  Overall: Injection 4 (0-28 days): number analyzed (Participants) | 11 | 12 | 11 | 10 | 11 | 7
  Overall: Injection 4 (0-28 days) | 48.000 [1.00 to 408.52] | 48.000 [4.00 to 604.77] | 48.000 [6.00 to 456.80] | 182.808 [8.00 to 629.07] | 30.067 [4.00 to 459.00] | 12.000 [6.00 to 48.00]
  Overall: Injection 6 (0-28 days): number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1
  Overall: Injection 6 (0-28 days) |  |  |  |  | 48.000 [48.00 to 48.00] | 48.000 [48.00 to 48.00]

21. Primary Outcome: Norbuprenorphine PK: Accumulation Index in Terms of Area Under the Curve (Rac(AUC))
Description: as for outcome 9
Time Frame: Days 1-28, 85-113
Population: PK population of participants with data at both timepoints
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Group 1 (8 mg) RBP-6000: 50 mg | Group 2 (12 mg) RBP-6000: 100 mg | Group 3 (24 mg) RBP-6000: 200 mg | Group 4 (8 mg) RBP-6000: 100 mg | Group 5 (14 mg) RBP-6000: 200 mg | Group 6 (8-24 mg) RBP-6000: 300 mg
Number analyzed (Participants) | 8 | 9 | 9 | 8 | 7 | 2
ratio | 1.071 (0.4044) | 1.924 (1.9274) | 1.147 (0.5899) | 1.709 (0.4088) | 1.711 (0.5931) | 1.247 (0.6737)

22. Primary Outcome: Norbuprenorphine PK: Accumulation Index in Terms of Maximum Observed Plasma Drug Concentration (Rac(Cmax))
Description: Accumulation index in terms of Cmax calculated as ratio of Cmax Injection 4/ Cmax Injection 1.
Time Frame: Days 1-28, 85-113
Population: PK population of participants with data at both timepoints
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Group 1 (8 mg) RBP-6000: 50 mg | Group 2 (12 mg) RBP-6000: 100 mg | Group 3 (24 mg) RBP-6000: 200 mg | Group 4 (8 mg) RBP-6000: 100 mg | Group 5 (14 mg) RBP-6000: 200 mg | Group 6 (8-24 mg) RBP-6000: 300 mg
Number analyzed (Participants) | 11 | 12 | 11 | 10 | 11 | 7
ratio | 0.300 (0.1294) | 0.697 (0.9077) | 0.272 (0.1131) | 0.548 (0.2978) | 0.445 (0.2231) | 0.730 (0.5830)

23. Primary Outcome: Norbuprenorphine PK: Area Under Plasma Concentration Time Curve From Time Zero Of Injection 4 and 6 (AUC0-∞)
Description: Area under plasma concentration time curve from time zero of Injection 4 extrapolated to infinity; calculated for Injection 4 and 6 (last injection) in subjects not participating in PET imaging sub-study only as:
  (AUC0-∞ was reported if the coefficient of determination R2 was at least 0.8 and the extrapolated area is less than 25%). A minimum of 5 data points was required. AUC up to the last measurable concentration (AUClast) was calculated by using the linear trapezoidal rule.
Time Frame: Days 85-113, 141-197
Population: PK population of participants whose data met requirements.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Group 1 (8 mg) RBP-6000: 50 mg | Group 2 (12 mg) RBP-6000: 100 mg | Group 3 (24 mg) RBP-6000: 200 mg | Group 4 (8 mg) RBP-6000: 100 mg | Group 5 (14 mg) RBP-6000: 200 mg | Group 6 (8-24 mg) RBP-6000: 300 mg
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 14
hr*ng/mL
  Overall: Injection 4 (0-28 days): number analyzed (Participants) | 3 | 4 | 2 | 0 | 1 | 0
  Overall: Injection 4 (0-28 days) | 499.733 (391.9606) | 1583.219 (1471.7341) | 639.892 (135.9113) |  | 1472.769 |
  Overall: Injection 6 (0-28 days): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Overall: Injection 6 (0-28 days) |  |  |  |  |  | 737.097

24. Primary Outcome: Norbuprenorphine PK: Terminal Phase Half Life (t1/2) Calculated For Injection 4
Description: as for outcome 13
Time Frame: Days 85-113, 141-197
Population: PK population of participants whose data met requirements.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Group 1 (8 mg) RBP-6000: 50 mg | Group 2 (12 mg) RBP-6000: 100 mg | Group 3 (24 mg) RBP-6000: 200 mg | Group 4 (8 mg) RBP-6000: 100 mg | Group 5 (14 mg) RBP-6000: 200 mg | Group 6 (8-24 mg) RBP-6000: 300 mg
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 14
hours
  Overall: Injection 4 (0-28 days): number analyzed (Participants) | 3 | 4 | 2 | 0 | 1 | 0
  Overall: Injection 4 (0-28 days) | 405.325 (47.4883) | 241.914 (114.8553) | 334.080 (48.0676) |  | 310.879 |
  Overall: Injection 6 (0-28 days): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Overall: Injection 6 (0-28 days) |  |  |  |  |  | 158.840

25. Secondary Outcome: Change From Baseline in the Clinical Opiate Withdrawal Scale (COWS) Prior to Injections 1, 2, 3, 4 and 6
Description: COWS is an 11-item instrument used to assess symptoms of opioid withdrawal (Wesson et al., 1999). The score is the sum of the responses for a total range of 0-48. The COWS is commonly used by clinicians treating patients with buprenorphine to monitor the severity of withdrawal. COWS scores below 5 are considered not indicative of withdrawal. Scores from 5 to 12 are considered mild withdrawal; from 13 to 24 moderate withdrawal; 25 to 36 moderate/severe withdrawal, and 37-48 severe withdrawal. Each participant was to be assessed by the same qualified and trained individuals throughout the course of the study as much as possible.
  Baseline was defined as the peak (maximum) value from screening to study Day -13 pre-SUBUTEX dose. The baseline score is reported as the mean of observed values. Other measurements were taken prior to dosing and reported as change from baseline values.
  Negative change from baseline values indicate a lessening of withdrawal symptoms.
Time Frame: Baseline (screening to Day -13), Days -1, 1, 29, 57, 85 141
Population: The pharmacodynamic (PD) population included subjects in Cohorts 1 - 6 who were dosed with RBP 6000 and had at least 1 post-dose value of the PD parameter.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 (8 mg) RBP-6000: 50 mg | Group 2 (12 mg) RBP-6000: 100 mg | Group 3 (24 mg) RBP-6000: 200 mg | Group 4 (8 mg) RBP-6000: 100 mg | Group 5 (14 mg) RBP-6000: 200 mg | Group 6 (8-24 mg) RBP-6000: 300 mg
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 14
units on a scale
  Baseline (observed values) | 17.6 (3.18) | 17.7 (3.22) | 20.4 (4.42) | 16.2 (2.91) | 17.9 (3.65) | 16.7 (2.33)
  Day -1 | -16.53 (3.335) | -16.33 (4.152) | -19.33 (4.670) | -15.50 (2.324) | -16.80 (3.986) | -15.93 (2.056)
  Day 1 | -16.67 (3.155) | -16.73 (3.788) | -19.27 (4.891) | -15.60 (2.720) | -16.87 (3.563) | -16.36 (2.341)
  Day 29: number analyzed (Participants) | 15 | 14 | 13 | 13 | 14 | 11
  Day 29 | -16.80 (2.908) | -16.79 (3.262) | -19.92 (4.663) | -15.77 (3.059) | -16.71 (3.989) | -16.91 (2.548)
  Day 57: number analyzed (Participants) | 12 | 13 | 11 | 12 | 13 | 10
  Day 57 | -17.75 (3.108) | -16.62 (3.776) | -18.91 (4.253) | -16.08 (2.937) | -17.62 (3.453) | -17.00 (2.449)
  Day 85: number analyzed (Participants) | 11 | 12 | 11 | 10 | 11 | 7
  Day 85 | -18.09 (3.015) | -17.08 (3.895) | -19.55 (4.059) | -16.10 (2.998) | -18.00 (3.873) | -16.00 (2.828)
  Day 141: number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 2
  Day 141 |  |  |  |  | -19.67 (4.041) | -18.00 (4.243)

26. Secondary Outcome: Change From Baseline in the Subjective Opiate Withdrawal Scale (SOWS) Prior to Injections 1, 2, 3, 4 and 6
Description: The Subjective Opiate Withdrawal Scale (SOWS) contains 16 symptoms whose intensity the participant rates on a scale of 0 (not at all) to 4 (extremely) for a full scale of 0 (no withdrawal symptoms) to 64 (extreme withdrawal symptoms).
  Baseline was defined as the peak (maximum) value from screening to study Day -13 pre-SUBUTEX dose. The baseline score is reported as the mean of observed values. Other measurements were taken prior to dosing and reported as change from baseline values.
  Negative change from baseline values indicate a lessening of withdrawal symptoms.
Time Frame: Baseline (screening to Day -13), Days -1, 1, 29, 57, 85 141
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 (8 mg) RBP-6000: 50 mg | Group 2 (12 mg) RBP-6000: 100 mg | Group 3 (24 mg) RBP-6000: 200 mg | Group 4 (8 mg) RBP-6000: 100 mg | Group 5 (14 mg) RBP-6000: 200 mg | Group 6 (8-24 mg) RBP-6000: 300 mg
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 14
units on a scale
  Baseline (observed values) | 40.2 (11.14) | 47.8 (14.65) | 45.1 (11.89) | 42.7 (13.80) | 42.1 (15.41) | 43.9 (16.20)
  Day -1 | -38.07 (11.145) | -45.20 (16.794) | -43.40 (12.385) | -40.67 (13.563) | -39.47 (16.048) | -42.71 (17.117)
  Day 1 | -38.73 (11.285) | -45.60 (16.106) | -43.47 (12.489) | -40.80 (13.624) | -39.67 (15.041) | -42.57 (16.603)
  Day 29: number analyzed (Participants) | 15 | 14 | 13 | 13 | 14 | 11
  Day 29 | -38.20 (12.616) | -45.64 (16.832) | -44.15 (11.689) | -40.62 (13.997) | -39.64 (15.979) | -46.00 (15.205)
  Day 57: number analyzed (Participants) | 12 | 14 | 11 | 12 | 13 | 10
  Day 57 | -39.50 (11.844) | -46.07 (16.717) | -43.09 (11.631) | -39.50 (13.945) | -38.85 (15.486) | -49.20 (12.770)
  Day 85: number analyzed (Participants) | 11 | 12 | 11 | 10 | 11 | 7
  Day 85 | -38.36 (11.595) | -45.58 (16.654) | -43.82 (11.763) | -41.60 (14.819) | -41.27 (15.691) | -51.71 (13.793)
  Day 141: number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 2
  Day 141 |  |  |  |  | -45.67 (5.132) | -59.50 (6.364)

27. Secondary Outcome: Change From Baseline in the Clinical Opioid Craving Visual Analog Scale (VAS) Total Score Prior to Injections 1, 2, 3, 4 and 6
Description: The Total Score was the sum of 10 questions regarding cravings each ranging from 0 (no craving) - 10 (extreme craving) for a total range from 0 (no cravings") to 100 ("most intense craving I have ever had").
  Baseline was defined as the peak (maximum) value from screening to study Day -13 pre-SUBUTEX dose. The baseline score is reported as the mean of observed values. Other measurements were taken prior to dosing and reported as change from baseline values.
  Negative change from baseline values indicate a lessening of craving symptoms.
Time Frame: Baseline (screening to Day -13), Days -1, 1, 29, 57, 85 141
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 (8 mg) RBP-6000: 50 mg | Group 2 (12 mg) RBP-6000: 100 mg | Group 3 (24 mg) RBP-6000: 200 mg | Group 4 (8 mg) RBP-6000: 100 mg | Group 5 (14 mg) RBP-6000: 200 mg | Group 6 (8-24 mg) RBP-6000: 300 mg
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 14
units on a scale
  Baseline (observed values) | 85.6 (9.98) | 89.7 (10.13) | 87.2 (10.41) | 86.0 (7.67) | 85.1 (12.64) | 87.4 (11.56)
  Day -1 | -84.00 (10.569) | -86.93 (14.255) | -84.53 (11.141) | -83.33 (8.449) | -82.07 (12.975) | -85.21 (11.088)
  Day 1 | -84.47 (10.569) | -88.20 (11.027) | -84.40 (11.451) | -83.73 (8.293) | -83.00 (12.689) | -85.36 (11.263)
  Day 29: number analyzed (Participants) | 15 | 14 | 13 | 13 | 14 | 11
  Day 29 | -81.73 (15.975) | -85.00 (12.247) | -85.31 (11.272) | -83.46 (8.771) | -82.36 (14.836) | -88.45 (10.377)
  Day 57: number analyzed (Participants) | 12 | 14 | 11 | 12 | 13 | 10
  Day 57 | -84.42 (11.437) | -86.64 (11.167) | -86.36 (11.792) | -82.08 (9.229) | -83.85 (13.459) | -88.10 (10.482)
  Day 85: number analyzed (Participants) | 11 | 12 | 11 | 10 | 11 | 7
  Day 85 | -84.91 (12.136) | -84.92 (13.507) | -86.55 (11.725) | -85.70 (6.848) | -89.27 (7.157) | -87.14 (11.668)
  Day 141: number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 2
  Day 141 |  |  |  |  | -85.33 (1.528) | -85.00 (4.243)

28. Secondary Outcome: Change From Baseline in the Clinical Global Impression Severity (CGI-S) Scale on Days 1, 7, 29, 57, 85 and 141
Description: The CGI-S is a 7-item scale completed by the clinician used to rate the severity of symptoms. The total range is 1 (normal, not at all ill) to 7 (most extremely ill).
  Baseline was defined as value from screening (Day -13). The baseline score is reported as the mean of observed values. Other measurements were taken prior to dosing (not applicable for Day 7) and reported as change from baseline values.
  Negative change from baseline values indicate a lessening of the severity of symptoms.
Time Frame: Baseline (screening Day -15), Days 1, 7, 29, 57, 85, 141
Population: The pharmacodynamic (PD) population included subjects in Cohorts 1 - 6 who were dosed with RBP 6000 and had at least 1 post-dose value of the PD parameter. One participant from Group 2 did not have a baseline evaluation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 (8 mg) RBP-6000: 50 mg | Group 2 (12 mg) RBP-6000: 100 mg | Group 3 (24 mg) RBP-6000: 200 mg | Group 4 (8 mg) RBP-6000: 100 mg | Group 5 (14 mg) RBP-6000: 200 mg | Group 6 (8-24 mg) RBP-6000: 300 mg
Number analyzed (Participants) | 15 | 14 | 15 | 15 | 15 | 14
units on a scale
  Baseline (observed values) | 4.3 (0.49) | 4.3 (0.61) | 4.4 (0.51) | 4.6 (0.51) | 4.7 (0.72) | 4.6 (0.51)
  Day 1: number analyzed (Participants) | 15 | 14 | 15 | 15 | 15 | 13
  Day 1 | 0.00 (0.000) | 0.00 (0.000) | 0.13 (0.352) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)
  Day 7: number analyzed (Participants) | 6 | 10 | 12 | 0 | 0 | 0
  Day 7 | -1.00 (1.095) | -0.50 (0.527) | -1.25 (0.965) |  |  |
  Day 29: number analyzed (Participants) | 15 | 14 | 13 | 13 | 14 | 11
  Day 29 | -1.40 (1.056) | -1.00 (1.038) | -1.23 (0.927) | -1.38 (0.961) | -1.64 (0.929) | -1.91 (1.044)
  Day 57: number analyzed (Participants) | 12 | 14 | 11 | 12 | 13 | 10
  Day 57 | -1.75 (1.055) | -1.29 (1.204) | -1.91 (1.221) | -1.83 (1.115) | -2.00 (1.000) | -2.50 (1.269)
  Day 85: number analyzed (Participants) | 11 | 12 | 11 | 10 | 11 | 7
  Day 85 | -1.82 (0.751) | -1.83 (1.115) | -2.18 (0.874) | -2.30 (1.160) | -2.64 (1.120) | -2.86 (1.345)
  Day 141: number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 2
  Day 141 |  |  |  |  | -3.00 (1.000) | -2.00 (2.828)

29. Secondary Outcome: Change From Baseline in the Clinical Global Impression Improvement (CGI-I) Scale on Days 7, 29, 57, 85 and 141
Description: The CGI-I is a 7-item scale completed by the clinician used to rate their impression of how much the participant has improved over a baseline state. The total range is 1 (very much improved) to 7 (very much worse).
  Baseline was defined as value from Day 1. The baseline score is reported as the mean of observed values. Other measurements were taken prior to dosing (not applicable for Day 7) and reported as change from baseline values.
  Negative change from baseline values indicate an improvement.
Time Frame: Baseline (Day 1), Days 7, 29, 57, 85, 141
Population: The pharmacodynamic (PD) population included subjects in Cohorts 1 - 6 who were dosed with RBP 6000 and had at least 1 post-dose value of the PD parameter. One participant from Group 6 did not have a baseline evaluation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 (8 mg) RBP-6000: 50 mg | Group 2 (12 mg) RBP-6000: 100 mg | Group 3 (24 mg) RBP-6000: 200 mg | Group 4 (8 mg) RBP-6000: 100 mg | Group 5 (14 mg) RBP-6000: 200 mg | Group 6 (8-24 mg) RBP-6000: 300 mg
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 13
units on a scale
  Baseline (observed values) | 4.0 (0.00) | 4.1 (0.26) | 4.0 (0.00) | 4.0 (0.00) | 4.0 (0.00) | 4.0 (0.00)
  Day 7: number analyzed (Participants) | 6 | 11 | 12 | 0 | 0 | 0
  Day 7 | -1.00 (1.095) | -0.73 (0.905) | -1.42 (1.084) |  |  |
  Day 29: number analyzed (Participants) | 15 | 14 | 13 | 13 | 14 | 11
  Day 29 | -1.67 (0.976) | -1.07 (1.072) | -1.77 (1.092) | -1.69 (0.947) | 02.07 (0.616) | -2.27 (1.191)
  Day 57: number analyzed (Participants) | 12 | 14 | 11 | 12 | 13 | 10
  Day 57 | -2.08 (0.793) | -1.79 (0.975) | -2.36 (0.809) | -2.17 (0.937) | -2.15 (0.801) | -2.40 (0.966)
  Day 85: number analyzed (Participants) | 11 | 12 | 11 | 10 | 11 | 7
  Day 85 | -2.18 (0.603) | -2.00 (0.953) | -2.73 (0.467) | -2.60 (0.699) | -2.73 (0.647) | -2.57 (0.787)
  Day 141: number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 2
  Day 141 |  |  |  |  | -2.67 (0.577) | -2.50 (0.707)

30. Secondary Outcome: Columbia Suicide Severity Rating Scale (C-SSRS): Severity
Description: The scale used in the C-SSRS is a continuous variable ranging from 0 (no suicidal ideation present) to 5 (active ideation with specific plan and intent). Only participants with suicidal ideation (scale of 1-5) are reported. 1=desire to be dead to 5=active ideation with specific plan and intent.
Time Frame: Screening (summary of lifetime), Screening (last 6 months), Day 65, Day 113, End of Study (up to day 365)
Population: PD population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 (8 mg) RBP-6000: 50 mg | Group 2 (12 mg) RBP-6000: 100 mg | Group 3 (24 mg) RBP-6000: 200 mg | Group 4 (8 mg) RBP-6000: 100 mg | Group 5 (14 mg) RBP-6000: 200 mg | Group 6 (8-24 mg) RBP-6000: 300 mg
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 14
units on a scale
  Screening (summary of lifetime): number analyzed (Participants) | 1 | 0 | 5 | 2 | 1 | 3
  Screening (summary of lifetime) | 1.0 |  | 1.8 (0.45) | 2.0 (1.41) | 1.0 | 1.3 (0.58)
  Screening (last 6 months): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Screening (last 6 months) |  |  |  |  |  | 1.0
  Day 65: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1
  Day 65 |  |  |  |  | 1.0 | 1.0
  Day 113: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  Day 113 |  | 1.0 |  |  |  |
  End of study: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0
  End of study |  |  | 5.0 |  |  |

31. Secondary Outcome: Percentage of Urine Drug Screen Samples Negative for Opioids
Description: Urine samples were screened for the following drugs:
  * opiates
  * cocaine
  * amphetamines
  * methadone
  * cannabinoids
  * barbiturates
  * buprenorphine. Buprenorphine was only included in the urine drug screen at screening and Day -14 to determine if the subject had used any buprenorphine-containing products prior to the start of SUBUTEX SL tablet dosing.
  * benzodiazepines
  * methamphetamine
  * phencyclidine
  Urine drug screens were run every day when the participant was an inpatient; every 2-3 days when the participant was an outpatient. Drug screens were run less often for those participants in the PET substudy.
Time Frame: Day 1 to End of Study (up to day 365)
Population: Safety population
Measure: Mean (Standard Deviation); unit: percentage of total urine drug samples
Arm/Group | Group 1 (8 mg) RBP-6000: 50 mg | Group 2 (12 mg) RBP-6000: 100 mg | Group 3 (24 mg) RBP-6000: 200 mg | Group 4 (8 mg) RBP-6000: 100 mg | Group 5 (14 mg) RBP-6000: 200 mg | Group 6 (8-24 mg) RBP-6000: 300 mg
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 14
percentage of total urine drug samples | 41.2 (32.89) | 42.0 (35.43) | 54.6 (23.98) | 49.9 (25.53) | 41.6 (27.68) | 64.9 (23.56)

ADVERSE EVENTS:
Time Frame: - Subutex Only Days -14 to Day -1 - Groups 1-4 (no PET substudy): Days -14 up to Day 141 - Groups 5-6 (including PET substudy): Days -14 up to Day 316
Groups:
- Group 5 (14 mg) RBP-6000: 200 mg: Participants are stabilized by day -5 on Subutex 14 mg. During the study, four subcutaneous (SC) injections containing RBP-6000 200 mg are given at 28 day intervals.
  Participants who reach Day 112 (and have received all 4 planned SC injections) have the option to participate in the Positron Emission Tomography (PET) Pilot substudy. In the PET Pilot sub-study participants remain on 200 mg SC injections at 28 day intervals for an additional 6-9 intervals until they complete an magnetic resonance imaging (MRI) and a PET scan and pharmacokinetic samples at week 1 and week 4 post injection.
Arm/Group | SUBUTEX Only | Group 1 (8 mg) RBP-6000: 50 mg | Group 2 (12 mg) RBP-6000: 100 mg | Group 3 (24 mg) RBP-6000: 200 mg | Group 4 (8 mg) RBP-6000: 100 mg | Group 5 (14 mg) RBP-6000: 200 mg | Group 6 (8-24 mg) RBP-6000: 300 mg
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/15 | 2/15 | 1/15 | 1/15 | 2/15 | 0/14
Other Adverse Events (participants affected / at risk) | 24/35 | 15/15 | 15/15 | 15/15 | 15/15 | 15/15 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SUBUTEX Only (N=35) | Group 1 (8 mg) RBP-6000: 50 mg (N=15) | Group 2 (12 mg) RBP-6000: 100 mg (N=15) | Group 3 (24 mg) RBP-6000: 200 mg (N=15) | Group 4 (8 mg) RBP-6000: 100 mg (N=15) | Group 5 (14 mg) RBP-6000: 200 mg (N=15) | Group 6 (8-24 mg) RBP-6000: 300 mg (N=14)
Lobar pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Personality disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pelvic inflammatory disease (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vaginitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SUBUTEX Only (N=35) | Group 1 (8 mg) RBP-6000: 50 mg (N=15) | Group 2 (12 mg) RBP-6000: 100 mg (N=15) | Group 3 (24 mg) RBP-6000: 200 mg (N=15) | Group 4 (8 mg) RBP-6000: 100 mg (N=15) | Group 5 (14 mg) RBP-6000: 200 mg (N=15) | Group 6 (8-24 mg) RBP-6000: 300 mg (N=14)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Leukoyctosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 1 | 1 | 0 | 2 | 2
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 3 | 2 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 2 | 4 | 5 | 4 | 7 | 5
Constipation (Gastrointestinal disorders) | 6 | 7 | 8 | 8 | 6 | 8 | 4
Nausea (Gastrointestinal disorders) | 2 | 1 | 2 | 3 | 1 | 6 | 2
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 2 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 1
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Faeces hard (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gingivitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Drug withdrawal syndrome (General disorders) | 12 | 9 | 11 | 13 | 13 | 14 | 7
Fatigue (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 3
Injection site pruritus (General disorders) | 0 | 1 | 2 | 2 | 0 | 0 | 3
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Facial pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Injection site pain (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Irritability (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza-like illness (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site dermatitis (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Injection site papule (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 2 | 0 | 2 | 0 | 0
Hepatic cyst (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Autoimmune disorder (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 4 | 5 | 5 | 3 | 2 | 6
Gastroenteritis (Infections and infestations) | 0 | 3 | 2 | 2 | 1 | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 2 | 2 | 0 | 1 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chlamydial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infective glossitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Perirectal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 2 | 2
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 3 | 1 | 2 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Testicular injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 2 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 2 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood creatinine phosphokinase increased (Investigations) | 0 | 2 | 2 | 0 | 0 | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 2 | 1 | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 1 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 2 | 1 | 0 | 0 | 0 | 1 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0 | 1 | 2 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 2 | 2 | 1 | 0
Weight increased (Investigations) | 0 | 1 | 1 | 2 | 0 | 1 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight fluctuation (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 9 | 7 | 6 | 3 | 4 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 3 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 8 | 7 | 6 | 9 | 7 | 9 | 7
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 0 | 2 | 0 | 2
Myoclonus (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Restless leg syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting in pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 6 | 9 | 5 | 2 | 4 | 8
Abnormal dreams (Psychiatric disorders) | 2 | 3 | 1 | 1 | 2 | 2 | 3
Insomnia (Psychiatric disorders) | 2 | 3 | 3 | 2 | 0 | 1 | 3
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intentional self-injury (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 3 | 1 | 2 | 1 | 0 | 0
Substance-induced mood disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Substance-induced psychotic disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 1 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 1 | 0 | 1 | 2
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 2 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 1 | 2 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Physical assault (Social circumstances) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 0
Bundle branch block right (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Orthostatic hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Proposed publications shall be submitted to Sponsor 30 days prior to submission for publication, and may be withheld for an additional period, up to 90 days, to allow Sponsor to file patent applications. If a multi-center publication isn't submitted for publication within 12 months of the conclusion of the Study at all sites, or is published in a shorter period, the results from the institution's site may be published individually.